CLINICAL TRIAL: NCT02445222
Title: Long Term Follow-Up of Patients Exposed to Lentiviral-Based CAR T-Cell Therapy
Brief Title: CAR-T Long Term Follow Up (LTFU) Study
Acronym: PAVO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCTL019A2205B; 2014-001673-14 (EudraCT Number)
Record Dates: First submitted 2015-05-01; First posted 2015-05-15 (Estimated); Last update posted 2025-10-28 (Actual); Status verified 2025-10

CONDITIONS: Long Term Safety of Patients Receiving CAR-T in an Eligible Clinical Trial or Managed Access Program

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Previously treated CAR-T patients (Other): Patients who previously were exposed to lentiviral-based CART cell therapy
  Interventions: Genetic: Previously treated CAR-T patients

INTERVENTIONS:
Genetic: Previously treated CAR-T patients — Lentiviral-based CAR-T cell therapy

SUMMARY:
Per Health Authorities guidelines for gene therapy medicinal products that utilize integrating vectors (e.g. lentiviral vectors), long term safety and efficacy follow up of treated patients is required. The purpose of this study is to monitor all patients exposed to CAR-T therapied for 15 years following their last CAR-T (e.g. CTL019) infusion to assess the risk of delayed adverse events (AEs), monitor for replication competent lentivirus (RCL) and assess long-term efficacy, including vector persistence.

DETAILED DESCRIPTION:
Patients are enrolled following completion or early discontinuation from a Novartis sponsored or supported study of CAR T-Cell treatment. Patients will be followed for 15 years post treatment from the last treatment. They will be monitored for safety and efficacy within the primary treatment protocols for the protocol defined duration. Patients can drop off treatment protocols at any time to enter this long term Follow up study. Patients discontinuing from the primary treatment protocols for any reason will be enrolled in this long term follow up (LTFU). This will allow collecting data on long term safety and efficacy (as applicable) as mandated by the health authorities of all patients treated with CAR-T therapy within the concept of a single protocol.

Collection of such long term effects of CAR-T cell therapy will help to further define the risk-benefit profile of CAR-T Therapies.

ELIGIBILITY:
Inclusion Criteria:

* All patients who have received a CAR-T therapy and completed or discontinued early from a Novartis sponsored treatment protocol that utilized CAR-T cells or from any CAR-T trial sponsored by the University of Pennsylvania with which Novartis has a contractual agreement to co-develop the CAR technology.
* Patients who have provided informed consent for the long term follow up study prior to their study participation .

Exclusion Criteria:

* There are no specific exclusion criteria for this study.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Start 2015-11-02 (Actual); Primary Completion 2036-02-22 (Estimated); Study Completion 2036-02-22 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with certain events (see description) | at M3 post treatment, M6, M9, M12 and then, every 6M up to year 5, yearly until year 15.
  The percentage of pts with listed categories: New secondary malignancies, new serious infection, new incidence of serious neurologic disorder, New incidence or exacerbation of a prior rheumatologic or other autoimmune disorder, New incidence of a hematologic disorder

SECONDARY OUTCOMES:
Percentage of patients with detectable CAR transgene levels in peripheral blood by q-PCR at pre- specified time points | at M3 post treatment, M6, M9, M12 and every 6M up to year 5, yearly until year 15.
Percentage of patients with detectable RCL by VSV-G | at M3 post treatment then M6, M9, M12 and every 6M up to year 5, yearly until year 15
Percentage of patients who relapse or progress among patients who had not relapsed or progressed at study entry/re-entry;Incidence of death | at M3 post treatment then M6, M9, M12 and every 6M up to year 5, yearly until year 15.
B- and T- lymphocyte count | at M3 post treatment then M6, M9, M12 and every 6M up to year 5, yearly until year 15.
Height and weight, Tanner staging, menstruation status | at M3 post treatment then M6, M12 and every year until year 15.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (102):
- United States (42):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - City of Hope National Medical Center, Duarte, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Emory University School of Medicine-Winship Cancer Institute, Atlanta, Georgia
  - Emory University School of Medicine/Winship Cancer Institute, Atlanta, Georgia
  - Childrens Healthcare of Atlanta, Atlanta, Georgia
  - Uni of Chi Medi Ctr Hema and Onco, Chicago, Illinois
  - University of Chicago Medical Center, Hematology & Oncology, Chicago, Illinois
  - University of Kansas Cancer Center SC, Westwood, Kansas
  - University of Kansas Cancer Center, Westwood, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Uni Of Michigan Health System, Ann Arbor, Michigan
  - University of Michigan Health System SC CTL019, Ann Arbor, Michigan
  - Wayne State University-Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Children s Mercy Hospital, Kansas City, Missouri
  - Children's Mercy Hospital SC, Kansas City, Missouri
  - Weill Cornell Medical College, New York, New York
  - Duke Unversity Medical Center SC - CTL019B2205J, Durham, North Carolina
  - Duke Unversity Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cinn Children Hosp Medical Center, Cincinnati, Ohio
  - Ohio ST Compr Cancer Ctr James Hosp, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - The Childrens Hosp of Philadelphia, Philadelphia, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - UTSW/Children's Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center SC, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Clinical Trials Office, Salt Lake City, Utah
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - University of Wisconsin Hospital, Madison, Wisconsin
- Australia (5):
  - Novartis Investigative Site, Camperdown, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Parkville, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
  - Novartis Investigative Site, Herston
- Austria (3):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Ghent, Belgium
- Canada (3):
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Beijing, China
- Novartis Investigative Site, Copenhagen, Denmark
- Novartis Investigative Site, Helsinki, Finland
- France (4):
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Villejuif
- Germany (9):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Frankfurt am Main, Hesse
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Chaïdári, Greece
- Novartis Investigative Site, Hong Kong, Hong Kong
- Israel (2):
  - Novartis Investigative Site, Ramat Gan
  - Novartis Investigative Site, Tel Aviv
- Italy (5):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Monza, MB
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Roma, RM
- Japan (5):
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sendai, Miyagi
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Kyoto
- Netherlands (2):
  - Novartis Investigative Site, Amsterdam, North Holland
  - Novartis Investigative Site, Utrecht
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Riyadh, Saudi Arabia
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Seoul, South Korea
- Spain (9):
  - Novartis Investigative Site, Esplugues, Barcelona
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Novartis Investigative Site, Taipei, Taiwan
- United Kingdom (2):
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, London

REFERENCES:
- [Derived] Maziarz RT, Bishop MR, Tam CS, Borchmann P, Worel N, McGuirk JP, Holte H, Waller EK, Jaglowski S, Andreadis C, Foley SR, Westin JR, Fleury I, Ho PJ, Mielke S, Teshima T, Janakiram M, Hsu J, Izutsu K, Kersten MJ, Ghosh M, Wagner-Johnston N, Kato K, Corradini P, Ma W, Han X, Nuortti M, Awasthi R, Mundt KE, Majdan M, Maier HJ, Jegerlehner A, Salles G, Schuster SJ. Five-Year Analysis of the JULIET Trial of Tisagenlecleucel in Patients With Relapsed/Refractory Large B-Cell Lymphoma. J Clin Oncol. 2026 Jan 10;44(2):86-91. doi: 10.1200/JCO-25-00507. Epub 2025 Nov 18. PMID 41252666